CLINICAL TRIAL: NCT01757093
Title: Evaluation of Oxygen Consumption and Energy Expenditure During Spontaneous Breathing Trial - A Randomized Crossover Controled Trial.
Brief Title: Evaluation of Oxygen Consumption and Energy Expenditure During Spontaneous Breathing Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Alessandra Fabiane Lago, ALESSANDRA FABIANE LAGO, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: AFL-0705
Record Dates: First submitted 2012-12-17; First posted 2012-12-28 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Respiratory Failure
Keywords: INDIRECT CALORIMETRY; MECHANICAL VENTILATION; WEANING VENTILATOR; AUTOMATIC TUBE COMPENSATION
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Automatic tube compensation plus CPAP (Experimental): The patients is going to undergo trials of spontaneous breathing with automatic tube compensation plus continuous positive airway pressure and later a trial with continuous positive airway pressure. During 30 minutes.
  Interventions: Device: Automatic Tube Compensation plus CPAP; Device: Continuous Positive Airway Pressure
- Continuous Positive Airway Pressure (Active Comparator): The patients is going to undergo a trial of spontaneous breathing with continuous positive airway pressure and later with automatic tube compensation plus continuous positive airway pressure, during 30 minutes each.
  Interventions: Device: Automatic Tube Compensation plus CPAP; Device: Continuous Positive Airway Pressure

INTERVENTIONS:
Device: Automatic Tube Compensation plus CPAP — SPONTANEOUS BREATHING TRIAL WITH AUTOMATIC TUBE COMPENSATION plus CPAP
  Other Names: ATC+CPAP
Device: Continuous Positive Airway Pressure — SPONTANEOUS BREATHING TRIAL WITH CPAP

SUMMARY:
The purpose of this study is to compare the oxygen consumption and energy expenditure during the spontaneous breathing trial.

DETAILED DESCRIPTION:
Patients is going to submit to the 2 spontaneous breathing trial ( Automatic tube compensation plus continuous positive airway pressure and continuous positive airway pressure without automatic tube compensation. The oxygen consumption and energy expenditure is going to measure during the spontaneous breathing trial by indirect calorimetry.

ELIGIBILITY:
Inclusion Criteria:

* IMPROVEMENT OR RESOLUTION OF THE UNDERLYING CAUSE OF DISEASE
* INTUBATED PATIENTS>24h
* PaO2 GREATER THAN 60 mmHg WITH FiO2 LESS THAN 40%
* PEEP=5 cmH2O

Exclusion Criteria:

* CARDIOVASCULAR INSTABILITY
* FEBRILE OR HYPOTHERMIA
* CHEST DRAINAGE
* RESPIRATORY RATE/TIDAL VOLUME RATIO GREATER THAN 105
* PREGNANCY
* FAIL IN THE SPONTANEOUS BREATHING TRIAL
* LEAKS IN THE CIRCUIT
* AGITATION
* NOT ACCEPT PARTICIPATE IN THE STUDY

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Measurement of oxygen consumption through indirect calorimetry. | The measurement is during the spontaneous breathing trial, 30 minutes.
  Measurements using indirect calorimetry for determination of oxygen consumption

SECONDARY OUTCOMES:
Measurement of energy expenditure through indirect calorimetry | The measurement is during the spontaneous breathing trial, 30 minutes.
  Measurement using indirect calorimetry for determination of energy expenditure.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Fa Lago, physiotherap, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital Das Clínicas Da Faculdade de Medicina de Ribeirão Preto -Universidade de São Paulo, Ribeirão Preto, São Paulo, Brazil